CLINICAL TRIAL: NCT03512743
Title: A Observational Study to Investigate the Relationship of Levels of Serum Ferritin, Bone Mineral Density and Bone Metabolism in Chinese Healthy Postmenopausal Women
Brief Title: Association of Serum Ferritin and Bone Mineral Density With Bone Metabolism in Chinese Healthy Postmenopausal Women
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, You-Jia Xu, Professor, Second Affiliated Hospital of Soochow University
Other Study IDs: Sencond Soochow U
Record Dates: First submitted 2018-04-15; First posted 2018-05-01 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Postmenopausal Osteoporosis; Iron Metabolism Disorders
Keywords: bone mineral density; bone turnover markers; ferritin
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Iron Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Large amounts of experimental and animal evidence have confirmed that iron accumulation is associated with bone loss. However, it is still lack of the clinical studies relating iron accumulation to bone loss, especially in the pathological conditions during our Chinese. In this study, the investigators aim to assess the association between the levels of serum ferritin and bone mineral density in Chinese healthy postmenopausal women.

DETAILED DESCRIPTION:
For the past few years, an increasing number of in vitro studies show the association of iron accumulation with bone loss, particularly in postmenopausal women. And body iron accumulation is accurately reflected by levels of serum ferritin in clinic. The levels of serum ferritin among healthy women are about 13-150μg/L, and we give a definition of iron accumulation when serum ferritin range from 500μg/L to 1000 μg/L. How will the bone mineral density change in iron accumulation? The investigators intend to perform this study to explore and establish the relational function and logical function between serum ferritin, bone mineral density and biochemical markers of bone metabolism in Chinese healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. healthy postmenopausal women
2. subjects aged 55 years or older

Exclusion Criteria:

1. subjects with acute or chronic inflammatory or infectious diseases
2. chronic liver or renal diseases
3. history of transfusion or iron therapy in the previous year
4. history of drug therapy such as bisphosphonates and glucocorticoids, which might have affected bone metabolism
5. subjects with hematonosis

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of postmenopausal women aged 55 years or older who shall undergone comprehensive routine health examinations at the Second Affiliated Hospital of Soochow University, and on whom BMD, serum ferritin concentrations and bone turnover markers will be measured.The visitors are usually healthy and receive extensive screening tests for early detection of malignancy, diabetes, osteoporosis, and other age-related disease.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
The concentrations of serum ferritin | 12 months
  Serum ferritin was assayed by an immunoradiometric method.

SECONDARY OUTCOMES:
Bone turnover markers(BTMs) | 12 months
  BTMs are classified as indices of either bone resorption or formation. During this study, we detect serum collagen type 1 cross-linked C-telopeptide(bone resorption marker) and Procollagen type I N-terminal propeptide(Bone formation marker).
Bone mineral density(BMD) | 12 months
  Bone mineral density (BMD) in femur and lumbar spine were measured by dual-energy X-ray absorptiometry.

CONTACTS AND LOCATIONS:
Overall Officials: Youjia Xu, Ph.D,M.D., Study Chair — Second Affiliated Hospital of Soochow University
Locations (1):
- Second Affiliated Hospital of Soochow University, Suzhou, Jiagnsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li GF, Pan YZ, Sirois P, Li K, Xu YJ. Iron homeostasis in osteoporosis and its clinical implications. Osteoporos Int. 2012 Oct;23(10):2403-8. doi: 10.1007/s00198-012-1982-1. Epub 2012 Apr 14. PMID 22525981
- [Background] Chon SJ, Choi YR, Roh YH, Yun BH, Cho S, Choi YS, Lee BS, Seo SK. Association between levels of serum ferritin and bone mineral density in Korean premenopausal and postmenopausal women: KNHANES 2008-2010. PLoS One. 2014 Dec 18;9(12):e114972. doi: 10.1371/journal.pone.0114972. eCollection 2014. PMID 25522357
- [Background] Jian J, Pelle E, Huang X. Iron and menopause: does increased iron affect the health of postmenopausal women? Antioxid Redox Signal. 2009 Dec;11(12):2939-43. doi: 10.1089/ars.2009.2576. PMID 19527179
- [Background] Xiao W, Beibei F, Guangsi S, Yu J, Wen Z, Xi H, Youjia X. Iron overload increases osteoclastogenesis and aggravates the effects of ovariectomy on bone mass. J Endocrinol. 2015 Sep;226(3):121-34. doi: 10.1530/JOE-14-0657. Epub 2015 Jun 26. PMID 26116610